CLINICAL TRIAL: NCT03682081
Title: Impact of Novel Rehabilitative Approaches for Dysphagia in Patients With Alzheimer's Disease and Related Dementias
Brief Title: Interventions for Patients With Alzheimer's Disease and Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0835; A534255 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); K76AG068590 (NIH); Protocol Version 5/21/2024 (Other: UW Madison)
Record Dates: First submitted 2018-08-20; First posted 2018-09-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dementia; Dysphagia; Alzheimer Disease
Keywords: Dementia; Dysphagia; Alzheimer's Disease; Treatment; Lingual Strengthening; Saliva substitute
MeSH Terms: conditions — Dementia; Deglutition Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Usual care (No Intervention): Usual care groups will receive standard swallowing interventions identified by the Speech-Language Pathologist as appropriate to treat the patient's dysphagia and common in clinical practice. Such treatment would likely consist of dietary (e.g., thickened liquids or pureed foods) or postural compensatory strategies (e.g., chin down posture while swallowing). No progressive lingual strengthening approaches or regimented salivary substitute protocols are utilized.
- Saliva Substitute Intervention (Experimental): Each patient-caregiver dyad will be provided with a commercially available gel-based saliva substitute, Biotene® Oral Balance Gel that will be applied to the oral cavity regularly for 8 weeks.
  Interventions: Device: Biotene Oral Balance Gel
- Lingual Strengthening Intervention (Experimental): Patient-caregiver dyads will be trained in the lingual strengthening protocol and patients will undergo this intervention for 8 weeks. Isometric tongue strengthening will be facilitated by the Iowa Oral Performance Instrument (IOPI) device.
  Interventions: Device: Isometric tongue strengthening facilitated by Iowa Oral Performance Instrument (IOPI)
- Saliva Substitute and Lingual Strengthening Intervention (Experimental): Each patient-caregiver dyad will be provided with a commercially available gel-based saliva substitute, Biotene® Oral Balance Gel that will be applied regularly to the oral cavity for 8 weeks. Each dyad will also be trained in the lingual strengthening protocol and will undergo this intervention for 8 weeks. Isometric tongue strengthening will be facilitated by the Iowa Oral Performance Instrument (IOPI) device.
  Interventions: Device: Isometric tongue strengthening facilitated by Iowa Oral Performance Instrument (IOPI); Device: Biotene Oral Balance Gel

INTERVENTIONS:
Device: Isometric tongue strengthening facilitated by Iowa Oral Performance Instrument (IOPI) — An air-filled pressure bulb is placed on the surface of the oral tongue and pressed against the hard palate during exercise. Each patient is given a target pressure value to aim for as determined by the baseline one repetition maximum (1RM) lingual pressures. During week one of the regimen, the target value of each repetition will be 60% of the 1RM. For the remaining seven weeks, the target value will be increased to 80% of the 1RM. At weeks three, five, and seven, the baseline will be re-measured by phone and the 80% target value re-calculated.
  Other Names: Tongue strengthening
  Arms: Lingual Strengthening Intervention; Saliva Substitute and Lingual Strengthening Intervention
Device: Biotene Oral Balance Gel — Participants will be instructed to apply an amount equivalent to about 1 cm of Biotene® Oral Balance Gel with a finger to the tongue and most intensely affected areas of the oral cavity three times a day after brushing their teeth for 8 weeks.
  Other Names: Saliva substitute
  Arms: Saliva Substitute Intervention; Saliva Substitute and Lingual Strengthening Intervention

SUMMARY:
The overall purpose of this project is to develop effective dysphagia rehabilitative interventions for patients with Alzheimer's Disease and related dementias at risk for pneumonia development.

DETAILED DESCRIPTION:
This proposal consists of a small, randomized clinical trial to determine the impact of two novel interventions on swallowing-related outcomes in patients with mild-moderate Alzheimer's Disease and Related Dementias (ADRD) and identify subgroups of patients most likely to benefit from these interventions. Patient-caregiver dyads will be randomized to lingual strengthening, saliva substitute use, a combination of the two, or only usual care. Saliva and swallowing-related outcomes will be collected at baseline and following the 8 week intervention period.

Consent and Randomization: Eligible dyads will be approached, consented and randomized at clinical care sites within University of Wisconsin Hospital and Clinics. Eligible participants' capacity to consent will determined by their primary clinical provider or team. Research staff will consent participant (or legally authorized representatives) prior to their swallow study. Each dyad will have equal chances of randomization to either usual care or one of the intervention arms plus usual care, with randomization stratified by the participant's dementia severity determined by the Clinical Dementia Rating (CDR) scale to ensure equal distribution of mild and moderate patients.

Baseline Assessment: Following randomization, the baseline assessment will be completed in tandem with the outpatient clinic visit. Staff will collect data on sociodemographics, comorbidities (using the Charlson comorbidity score approach) and medications (including anticholinergics and neuroleptics). The Montreal Cognitive Assessment (MoCA) will be administered at this time. Oral health status will be graded using the Brief Oral Health Status Examination, a valid and reliable scoring instrument developed for non-dental health care providers in long term care. Dentition will be characterized by the number of posterior occlusal pairs of teeth and denture use. Smoking history and active use during the study will be recorded.

Usual Care: Usual care group participants will receive standard swallowing interventions as recommended by the clinical Speech-Language Pathologist. Such treatment would likely consist of dietary (e.g., thickened liquids or pureed foods) or postural compensatory strategies (e.g., chin down posture while swallowing). All patient participants in intervention groups will also receive usual care, as indicated per their primary clinical team.

Interventions:

Saliva substitute: Each patient-caregiver dyad will be provided with a commercially available gel-based saliva substitute, Biotene® Oral Balance Gel. Participants will be instructed to apply an amount equivalent to about 1 cm of gel with a finger to the tongue and most intensely affected areas of the oral cavity three times a day for 8 weeks. Caregivers will be trained in how to assist the patient with application and support will be provided through follow-up phone calls.

Lingual strengthening intervention: Device training for dyads assigned to lingual strengthening will occur following randomization during the research visit. Isometric tongue strengthening will be completed using the Iowa Oral Performance Instrument (IOPI) over an 8-week program. An air-filled pressure bulb is placed on the surface of the oral tongue and pressed against the hard palate during exercise. Each patient is given a target pressure value to aim for as determined by the baseline one repetition maximum (1RM) lingual pressures. During week one of the regimen, the target value of each repetition will be 60% of the 1RM. For the remaining seven weeks, the target value will be increased to 80% of the 1RM. At weeks three, five, and seven, the baseline will be re-measured by phone and the 80% target value re-calculated. The final assessment point will be after completion of lingual strengthening. Training will be provided to both participants and caregivers on the device and lingual strengthening protocol and support will be provided to dyads through follow-up phone calls.

ELIGIBILITY:
Inclusion criteria (patients):

* Age 50-99
* English speaking
* Diagnosis of dementia or cognitive impairment or memory loss
* Clinical Dementia Rating (CDR) scale score between 0.5 and 2.0
* Actively involved caregiver
* Resides at home, assisted living facility, or long-term care facility

Inclusion criteria (caregivers)

* English speaking
* Age 18 and older
* Contact with patient at least 1 time a week
* Has access to a working telephone

Exclusion criteria (patients):

* Dementia due to cerebrovascular disease as primary cause
* History of head and neck cancer or other structural deformity that can affect swallowing
* Allergy to barium
* Currently breastfeed or pregnant or planning to become pregnant

Exclusion criteria (caregivers):

* Lacks ability to give consent

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Pharyngeal residue measured with the Normalized Residue Ratio Scale (NRRS) | Baseline, Post-treatment at approximately 8 weeks
  Pixel-based measure of post-swallow pharyngeal barium residue as observed on a videofluoroscopic swallow study captured at 30 frames per second. This measure will represent the amount of pharyngeal residue as it relates to the distance between cervical vertebrae 2 and 4 which serve as an anatomical scalar. A higher value represents more pharyngeal residue which is a worse outcome.

SECONDARY OUTCOMES:
Change in Modified Barium Swallow Impairment Profile (MBSImP) Overall Impairment Scores | Baseline, Post-treatment at approximately 8 weeks
  Assessment of swallow function is completed though examination of 17 physiologic components requisite for the execution of normal swallowing. MBSImP includes an operationally defined scoring metric for each component that is applied to accurately describe and quantify progressing levels of impairment. Total possible range of scores is 0-62 with higher scores indicative of increased impairment.
Change in Penetration-Aspiration Scale Scores | Baseline, Post-treatment at approximately 8 weeks
  The penetration-aspiration scale, a validated scale used to measure the severity of airway invasion with swallowing, will be used with recordings of videofluoroscopic swallow studies. This is an 8-point scale with no airway invasion represented by a score of 1 and aspiration with no response represented by a score of 8. A higher score represents a worse outcome.
Change in Lingual strength-maximal isometric lingual pressures | Baseline, Post-treatment at approximately 8 weeks
  Maximum lingual pressures will be measured at the anterior and posterior locations of the tongue using the Iowa Oral Performance Instrument (IOPI). A higher value represents greater lingual pressure generation which is a better outcome.
Change in Functional Oral Intake Scale | Baseline, Post-treatment at approximately 8 weeks
  This is a validated scale used the quantify the level of oral versus nonoral intake as well as any dietary modifications needed. A score of 1 represents no oral intake with complete dependence on a feeding tube while a score of 7 represents total oral intake with no diet modifications. A higher score represents a better outcome.
Change in Swallowing Quality of Life Questionnaire | Baseline, Post-treatment at approximately 8 weeks.
  The Swal-QOL is a validated questionnaire focused on swallowing-related quality of life. It comprises 10 multi-item scales, 2 general scales, and a 14-item symptom battery. Total possible range of scores is 0-100, higher scores represent better quality of life.
Change in Zarit Burden Interview | Baseline, Post-treatment at approximately 8 weeks
  The Zarit Caregiver Burden Scale is used as a measure of caregiver psychological stress. The scores across all 22 items are summed and the range for the total score is from 0-88 with higher scores indicating greater burden (a worse outcome).
Change in Pneumonia diagnoses | Post-enrollment at approximately days 7, 14, 28, 42, 56, 90, and 180
  As an exploratory outcome, we will review the electronic health record for all pneumonia diagnoses (ICD-10 codes)for 180 days after enrollment in the study. A decrease in the number of pneumonia diagnoses represents improvement.
Change in Salivary Production Rates | Baseline, Post-treatment at approximately 8 weeks
  Saliva production will be quantified through weighing collection tubes before and after unstimulated and stimulated saliva collection. A higher saliva weight represents a greater salivary flow rate and more saliva production.
Change in Residual Mucosal Saliva (RMS) | Baseline, Post-treatment at approximately 8 weeks
  RMS correlates with hyposalivation and dryness perception, will be collected from the anterior hard palate (AHP), anterior tongue (AT), and lower labial (LL) surfaces using SialoPaper strips (Oraflow Inc., Smithtown, NY, USA). These strips will be applied for 10 seconds and measured using Periotron device (Oraflow Inc.).
Change in Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) scores | Baseline, Post-treatment at approximately 8 weeks
  Assessment of swallow function is completed though analysis of videofluoroscopic images for swallowing safety and efficiency with the DIGEST tool. This is a validated method for identifying and rating penetration, aspiration, and residue, resulting in an overall score. DIGEST scores combine an evaluation of individual swallows to determine a safety grade of 0-4 with an efficiency grade of 0-4 to determine an overall DIGEST grade of 0 (no impairment) to 4 (profound impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Rogus-Pulia, PhD, CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogus-Pulia N, Malandraki GA, Johnson S, & Robbins J. (2015). Understanding Dysphagia in dementia: The present and the future. Current Physical Medicine and Rehabilitation Reports, 3(1), 86-97.
- [Background] Foley NC, Affoo RH, Martin RE. A systematic review and meta-analysis examining pneumonia-associated mortality in dementia. Dement Geriatr Cogn Disord. 2015;39(1-2):52-67. doi: 10.1159/000367783. Epub 2014 Oct 22. PMID 25342272
- [Background] Alagiakrishnan K, Bhanji RA, Kurian M. Evaluation and management of oropharyngeal dysphagia in different types of dementia: a systematic review. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):1-9. doi: 10.1016/j.archger.2012.04.011. Epub 2012 May 19. PMID 22608838
- [Background] Kuroda Y. Factors associated with the level of oral intake in hospitalized older adults with dysphagia: The importance of mental activity. Clin Nutr ESPEN. 2016 Jun;13:e52-e54. doi: 10.1016/j.clnesp.2016.03.001. Epub 2016 Mar 27. PMID 28531569
- [Background] Riviere S, Gillette-Guyonnet S, Andrieu S, Nourhashemi F, Lauque S, Cantet C, Salva A, Frisoni G, Vellas B. Cognitive function and caregiver burden: predictive factors for eating behaviour disorders in Alzheimer's disease. Int J Geriatr Psychiatry. 2002 Oct;17(10):950-5. doi: 10.1002/gps.724. PMID 12325056
- [Background] Brunnstrom HR, Englund EM. Cause of death in patients with dementia disorders. Eur J Neurol. 2009 Apr;16(4):488-92. doi: 10.1111/j.1468-1331.2008.02503.x. PMID 19170740
- [Background] Wada H, Nakajoh K, Satoh-Nakagawa T, Suzuki T, Ohrui T, Arai H, Sasaki H. Risk factors of aspiration pneumonia in Alzheimer's disease patients. Gerontology. 2001 Sep-Oct;47(5):271-6. doi: 10.1159/000052811. PMID 11490146
- [Background] Milte R, Shulver W, Killington M, Bradley C, Miller M, Crotty M. Struggling to maintain individuality - Describing the experience of food in nursing homes for people with dementia. Arch Gerontol Geriatr. 2017 Sep;72:52-58. doi: 10.1016/j.archger.2017.05.002. Epub 2017 May 17. PMID 28552702
- [Background] Horner J, Alberts MJ, Dawson DV, Cook GM. Swallowing in Alzheimer's disease. Alzheimer Dis Assoc Disord. 1994 Fall;8(3):177-89. doi: 10.1097/00002093-199408030-00004. PMID 7986487
- [Background] Volicer L, Seltzer B, Rheaume Y, Karner J, Glennon M, Riley ME, Crino P. Eating difficulties in patients with probable dementia of the Alzheimer type. J Geriatr Psychiatry Neurol. 1989 Oct-Dec;2(4):188-95. doi: 10.1177/089198878900200404. PMID 2483945
- [Background] Easterling CS, Robbins E. Dementia and dysphagia. Geriatr Nurs. 2008 Jul-Aug;29(4):275-85. doi: 10.1016/j.gerinurse.2007.10.015. PMID 18694703
- [Background] Correia Sde M, Morillo LS, Jacob Filho W, Mansur LL. Swallowing in moderate and severe phases of Alzheimer's disease. Arq Neuropsiquiatr. 2010 Dec;68(6):855-61. doi: 10.1590/s0004-282x2010000600005. PMID 21243241
- [Background] Secil Y, Arici S, Incesu TK, Gurgor N, Beckmann Y, Ertekin C. Dysphagia in Alzheimer's disease. Neurophysiol Clin. 2016 Jun;46(3):171-8. doi: 10.1016/j.neucli.2015.12.007. Epub 2016 May 11. PMID 26924307
- [Background] Sakai K, Hirano H, Watanabe Y, Tohara H, Sato E, Sato K, Katakura A. An examination of factors related to aspiration and silent aspiration in older adults requiring long-term care in rural Japan. J Oral Rehabil. 2016 Feb;43(2):103-10. doi: 10.1111/joor.12349. Epub 2015 Oct 3. PMID 26432521
- [Background] Logemann JA, Gensler G, Robbins J, Lindblad AS, Brandt D, Hind JA, Kosek S, Dikeman K, Kazandjian M, Gramigna GD, Lundy D, McGarvey-Toler S, Miller Gardner PJ. A randomized study of three interventions for aspiration of thin liquids in patients with dementia or Parkinson's disease. J Speech Lang Hear Res. 2008 Feb;51(1):173-83. doi: 10.1044/1092-4388(2008/013). PMID 18230864
- [Background] Priefer BA, Robbins J. Eating changes in mild-stage Alzheimer's disease: a pilot study. Dysphagia. 1997 Fall;12(4):212-21. doi: 10.1007/PL00009539. PMID 9294942
- [Background] Humbert IA, McLaren DG, Kosmatka K, Fitzgerald M, Johnson S, Porcaro E, Kays S, Umoh EO, Robbins J. Early deficits in cortical control of swallowing in Alzheimer's disease. J Alzheimers Dis. 2010;19(4):1185-97. doi: 10.3233/JAD-2010-1316. PMID 20308785
- [Background] Campbell-Taylor I. Contribution of Alzheimer disease to mortality in the United States. Neurology. 2014 Sep 30;83(14):1302. doi: 10.1212/01.wnl.0000455099.43083.c6. No abstract available. PMID 25267987
- [Background] Paranji S, Paranji N, Wright S, Chandra S. A Nationwide Study of the Impact of Dysphagia on Hospital Outcomes Among Patients With Dementia. Am J Alzheimers Dis Other Demen. 2017 Feb;32(1):5-11. doi: 10.1177/1533317516673464. Epub 2016 Nov 9. PMID 27821563
- [Background] Favaro-Moreira NC, Krausch-Hofmann S, Matthys C, Vereecken C, Vanhauwaert E, Declercq A, Bekkering GE, Duyck J. Risk Factors for Malnutrition in Older Adults: A Systematic Review of the Literature Based on Longitudinal Data. Adv Nutr. 2016 May 16;7(3):507-22. doi: 10.3945/an.115.011254. Print 2016 May. PMID 27184278
- [Background] Lindroos E, Saarela RK, Soini H, Muurinen S, Suominen MH, Pitkala KH. Caregiver-reported swallowing difficulties, malnutrition, and mortality among older people in assisted living facilities. J Nutr Health Aging. 2014 Jul;18(7):718-22. doi: 10.1007/s12603-014-0506-4. PMID 25226112
- [Background] Nicosia MA, Hind JA, Roecker EB, Carnes M, Doyle J, Dengel GA, Robbins J. Age effects on the temporal evolution of isometric and swallowing pressure. J Gerontol A Biol Sci Med Sci. 2000 Nov;55(11):M634-40. doi: 10.1093/gerona/55.11.m634. PMID 11078092
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Background] Tolea MI, Galvin JE. Sarcopenia and impairment in cognitive and physical performance. Clin Interv Aging. 2015 Mar 30;10:663-71. doi: 10.2147/CIA.S76275. eCollection 2015. PMID 25878493
- [Background] FastStats - Alzheimers Disease. https://www.cdc.gov/nchs/fastats/alzheimers.htm. Accessed February 11, 2017.
- [Background] Namasivayam AM, Steele CM, Keller H. The effect of tongue strength on meal consumption in long term care. Clin Nutr. 2016 Oct;35(5):1078-83. doi: 10.1016/j.clnu.2015.08.001. Epub 2015 Aug 19. PMID 26321499
- [Background] Molfenter SM, Steele CM. The relationship between residue and aspiration on the subsequent swallow: an application of the normalized residue ratio scale. Dysphagia. 2013 Dec;28(4):494-500. doi: 10.1007/s00455-013-9459-8. Epub 2013 Mar 5. PMID 23460344
- [Background] Butler SG, Stuart A, Leng X, Wilhelm E, Rees C, Williamson J, Kritchevsky SB. The relationship of aspiration status with tongue and handgrip strength in healthy older adults. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):452-8. doi: 10.1093/gerona/glq234. Epub 2011 Feb 7. PMID 21300744
- [Background] Ship JA, DeCarli C, Friedland RP, Baum BJ. Diminished submandibular salivary flow in dementia of the Alzheimer type. J Gerontol. 1990 Mar;45(2):M61-6. doi: 10.1093/geronj/45.2.m61. PMID 2313044
- [Background] Affoo RH, Foley N, Garrick R, Siqueira WL, Martin RE. Meta-Analysis of Salivary Flow Rates in Young and Older Adults. J Am Geriatr Soc. 2015 Oct;63(10):2142-51. doi: 10.1111/jgs.13652. Epub 2015 Oct 12. PMID 26456531
- [Background] Borson S, Lampe T, Raskind M, Veith R, Morely J, Coe R, et al. (1992). Autonomic nervous system dysfunction in Alzheimer's disease: Implications for pathophysiology and treatment. Memory Function in Aging and Age-Related Disorders. New York: Springer Verlag, 175-189.
- [Background] Affoo RH, Foley N, Rosenbek J, Kevin Shoemaker J, Martin RE. Swallowing dysfunction and autonomic nervous system dysfunction in Alzheimer's disease: a scoping review of the evidence. J Am Geriatr Soc. 2013 Dec;61(12):2203-2213. doi: 10.1111/jgs.12553. PMID 24329892
- [Background] van der Bilt A, Engelen L, Abbink J, Pereira LJ. Effects of adding fluids to solid foods on muscle activity and number of chewing cycles. Eur J Oral Sci. 2007 Jun;115(3):198-205. doi: 10.1111/j.1600-0722.2007.00448.x. PMID 17587295
- [Background] Engelen L, van den Keybus PA, de Wijk RA, Veerman EC, Amerongen AV, Bosman F, Prinz JF, van der Bilt A. The effect of saliva composition on texture perception of semi-solids. Arch Oral Biol. 2007 Jun;52(6):518-25. doi: 10.1016/j.archoralbio.2006.11.007. Epub 2006 Dec 18. PMID 17178098
- [Background] Loesche WJ, Bromberg J, Terpenning MS, Bretz WA, Dominguez BL, Grossman NS, Langmore SE. Xerostomia, xerogenic medications and food avoidances in selected geriatric groups. J Am Geriatr Soc. 1995 Apr;43(4):401-7. doi: 10.1111/j.1532-5415.1995.tb05815.x. PMID 7706631
- [Background] Rogus-Pulia N, Robbins J. Approaches to the rehabilitation of dysphagia in acute poststroke patients. Semin Speech Lang. 2013 Aug;34(3):154-69. doi: 10.1055/s-0033-1358368. Epub 2013 Oct 28. PMID 24166190
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Behrman S, Chouliaras L, Ebmeier KP. Considering the senses in the diagnosis and management of dementia. Maturitas. 2014 Apr;77(4):305-10. doi: 10.1016/j.maturitas.2014.01.003. Epub 2014 Jan 18. PMID 24495787
- [Background] Aliani M, Udenigwe CC, Girgih AT, Pownall TL, Bugera JL, Eskin MN. Aroma and taste perceptions with Alzheimer disease and stroke. Crit Rev Food Sci Nutr. 2013;53(7):760-9. doi: 10.1080/10408398.2011.559557. PMID 23638935
- [Background] Roque M, Salva A, Vellas B. Malnutrition in community-dwelling adults with dementia (NutriAlz Trial). J Nutr Health Aging. 2013 Apr;17(4):295-9. doi: 10.1007/s12603-012-0401-9. PMID 23538648
- [Background] Colodny N. Dysphagic independent feeders' justifications for noncompliance with recommendations by a speech-language pathologist. Am J Speech Lang Pathol. 2005 Feb;14(1):61-70. doi: 10.1044/1058-0360(2005/008). PMID 15962847
- [Background] Robbins J, Gensler G, Hind J, Logemann JA, Lindblad AS, Brandt D, Baum H, Lilienfeld D, Kosek S, Lundy D, Dikeman K, Kazandjian M, Gramigna GD, McGarvey-Toler S, Miller Gardner PJ. Comparison of 2 interventions for liquid aspiration on pneumonia incidence: a randomized trial. Ann Intern Med. 2008 Apr 1;148(7):509-18. doi: 10.7326/0003-4819-148-7-200804010-00007. PMID 18378947
- [Background] van Halteren-van Tilborg IA, Scherder EJ, Hulstijn W. Motor-skill learning in Alzheimer's disease: a review with an eye to the clinical practice. Neuropsychol Rev. 2007 Sep;17(3):203-12. doi: 10.1007/s11065-007-9030-1. PMID 17680369
- [Background] Hauer K, Ullrich P, Dutzi I, Beurskens R, Kern S, Bauer J, Schwenk M. Effects of Standardized Home Training in Patients with Cognitive Impairment following Geriatric Rehabilitation: A Randomized Controlled Pilot Study. Gerontology. 2017;63(6):495-506. doi: 10.1159/000478263. Epub 2017 Aug 17. PMID 28813696
- [Background] Zieschang T, Schwenk M, Oster P, Hauer K. Sustainability of motor training effects in older people with dementia. J Alzheimers Dis. 2013;34(1):191-202. doi: 10.3233/JAD-120814. PMID 23202438
- [Background] Morris JK, Vidoni ED, Johnson DK, Van Sciver A, Mahnken JD, Honea RA, Wilkins HM, Brooks WM, Billinger SA, Swerdlow RH, Burns JM. Aerobic exercise for Alzheimer's disease: A randomized controlled pilot trial. PLoS One. 2017 Feb 10;12(2):e0170547. doi: 10.1371/journal.pone.0170547. eCollection 2017. PMID 28187125
- [Background] Fiatarone MA, Marks EC, Ryan ND, Meredith CN, Lipsitz LA, Evans WJ. High-intensity strength training in nonagenarians. Effects on skeletal muscle. JAMA. 1990 Jun 13;263(22):3029-34. PMID 2342214
- [Background] Robbins J. Upper aerodigestive tract neurofunctional mechanisms: lifelong evolution and exercise. Head Neck. 2011 Oct;33 Suppl 1(0 1):S30-6. doi: 10.1002/hed.21902. Epub 2011 Sep 9. PMID 21910155
- [Background] Juan J, Hind J, Jones C, McCulloch T, Gangnon R, Robbins J. Case study: application of isometric progressive resistance oropharyngeal therapy using the Madison Oral Strengthening Therapeutic device. Top Stroke Rehabil. 2013 Sep-Oct;20(5):450-70. doi: 10.1310/tsr2005-450. PMID 24091287
- [Background] Robison R. (2015). The Impact of Lingual Resistance Training in Two Individuals with Amyotrophic Lateral Sclerosis: A Case Series. University of South Florida Scholar Commons.
- [Background] Maguire A, Rugg-Gunn AJ. Xylitol and caries prevention--is it a magic bullet? Br Dent J. 2003 Apr 26;194(8):429-36. doi: 10.1038/sj.bdj.4810022. No abstract available. PMID 12778091
- [Background] Burgess J, Lee P. XyliMelts time-release adhering discs for night-time oral dryness. Int J Dent Hyg. 2012 May;10(2):118-21. doi: 10.1111/j.1601-5037.2011.00532.x. Epub 2011 Oct 31. PMID 22040224
- [Background] Ship JA, McCutcheon JA, Spivakovsky S, Kerr AR. Safety and effectiveness of topical dry mouth products containing olive oil, betaine, and xylitol in reducing xerostomia for polypharmacy-induced dry mouth. J Oral Rehabil. 2007 Oct;34(10):724-32. doi: 10.1111/j.1365-2842.2006.01718.x. PMID 17824884
- [Background] Gil-Montoya JA, Guardia-Lopez I, Gonzalez-Moles MA. Evaluation of the clinical efficacy of a mouthwash and oral gel containing the antimicrobial proteins lactoperoxidase, lysozyme and lactoferrin in elderly patients with dry mouth--a pilot study. Gerodontology. 2008 Mar;25(1):3-9. doi: 10.1111/j.1741-2358.2007.00197.x. Epub 2008 Jan 13. PMID 18194332
- [Background] Montine TJ, Koroshetz WJ, Babcock D, Dickson DW, Galpern WR, Glymour MM, Greenberg SM, Hutton ML, Knopman DS, Kuzmichev AN, Manly JJ, Marder KS, Miller BL, Phelps CH, Seeley WW, Sieber BA, Silverberg NB, Sutherland M, Torborg CL, Waddy SP, Zlokovic BV, Corriveau RA; ADRD 2013 Conference Organizing Committee. Recommendations of the Alzheimer's disease-related dementias conference. Neurology. 2014 Aug 26;83(9):851-60. doi: 10.1212/WNL.0000000000000733. Epub 2014 Jul 30. PMID 25080517
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Hind JA, Nicosia MA, Roecker EB, Carnes ML, Robbins J. Comparison of effortful and noneffortful swallows in healthy middle-aged and older adults. Arch Phys Med Rehabil. 2001 Dec;82(12):1661-5. doi: 10.1053/apmr.2001.28006. PMID 11733879
- [Background] Robbins J, Gangnon RE, Theis SM, Kays SA, Hewitt AL, Hind JA. The effects of lingual exercise on swallowing in older adults. J Am Geriatr Soc. 2005 Sep;53(9):1483-9. doi: 10.1111/j.1532-5415.2005.53467.x. PMID 16137276
- [Background] Rogus-Pulia N, Rusche N, Hind JA, Zielinski J, Gangnon R, Safdar N, Robbins J. Effects of Device-Facilitated Isometric Progressive Resistance Oropharyngeal Therapy on Swallowing and Health-Related Outcomes in Older Adults with Dysphagia. J Am Geriatr Soc. 2016 Feb;64(2):417-24. doi: 10.1111/jgs.13933. Epub 2016 Jan 25. PMID 26804715
- [Background] Christa Maree Stephan B, Minett T, Pagett E, Siervo M, Brayne C, McKeith IG. Diagnosing Mild Cognitive Impairment (MCI) in clinical trials: a systematic review. BMJ Open. 2013 Feb 4;3(2):e001909. doi: 10.1136/bmjopen-2012-001909. Print 2013. PMID 23386579
- [Background] Winchester J, & Winchester C. (2015). Cognitive dysphagia and effectively managing the five systems. Perspectives of the American Speech-Language-Hearing Association Special Interest Groups, 20.
- [Background] Rogus-Pulia NM, Gangnon R, Kind A, Connor NP, Asthana S. A Pilot Study of Perceived Mouth Dryness, Perceived Swallowing Effort, and Saliva Substitute Effects in Healthy Adults Across the Age Range. Dysphagia. 2018 Apr;33(2):200-205. doi: 10.1007/s00455-017-9846-7. Epub 2017 Sep 6. PMID 28879557
- [Background] Zussman E, Yarin AL, Nagler RM. Age- and flow-dependency of salivary viscoelasticity. J Dent Res. 2007 Mar;86(3):281-5. doi: 10.1177/154405910708600316. PMID 17314263
- [Background] Rudney JD, Ji Z, Larson CJ. The prediction of saliva swallowing frequency in humans from estimates of salivary flow rate and the volume of saliva swallowed. Arch Oral Biol. 1995 Jun;40(6):507-12. doi: 10.1016/0003-9969(95)00004-9. PMID 7677595
- [Background] Nogueira D, Reis E. Swallowing disorders in nursing home residents: how can the problem be explained? Clin Interv Aging. 2013;8:221-7. doi: 10.2147/CIA.S39452. Epub 2013 Feb 19. PMID 23449951
- [Background] Troche MS, Okun MS, Rosenbek JC, Altmann LJ, Sapienza CM. Attentional resource allocation and swallowing safety in Parkinson's disease: a dual task study. Parkinsonism Relat Disord. 2014 Apr;20(4):439-43. doi: 10.1016/j.parkreldis.2013.12.011. Epub 2014 Jan 8. PMID 24444532
- [Background] Kim JS, Youn J, Suh MK, Kim TE, Chin J, Park S, Cho JW. Cognitive and Motor Aspects of Parkinson's Disease Associated with Dysphagia. Can J Neurol Sci. 2015 Nov;42(6):395-400. doi: 10.1017/cjn.2015.304. PMID 26551089
- [Background] Leder SB, Suiter DM, Lisitano Warner H. Answering orientation questions and following single-step verbal commands: effect on aspiration status. Dysphagia. 2009 Sep;24(3):290-5. doi: 10.1007/s00455-008-9204-x. Epub 2009 Mar 5. PMID 19263106
- [Background] Keesman M, Aarts H, Vermeent S, Hafner M, Papies EK. Consumption Simulations Induce Salivation to Food Cues. PLoS One. 2016 Nov 7;11(11):e0165449. doi: 10.1371/journal.pone.0165449. eCollection 2016. PMID 27820842
- [Background] Langmore SE, Terpenning MS, Schork A, Chen Y, Murray JT, Lopatin D, Loesche WJ. Predictors of aspiration pneumonia: how important is dysphagia? Dysphagia. 1998 Spring;13(2):69-81. doi: 10.1007/PL00009559. PMID 9513300
- [Background] Furuta M, Komiya-Nonaka M, Akifusa S, Shimazaki Y, Adachi M, Kinoshita T, Kikutani T, Yamashita Y. Interrelationship of oral health status, swallowing function, nutritional status, and cognitive ability with activities of daily living in Japanese elderly people receiving home care services due to physical disabilities. Community Dent Oral Epidemiol. 2013 Apr;41(2):173-81. doi: 10.1111/cdoe.12000. Epub 2012 Aug 30. PMID 22934613
- [Background] Scully C. Drug effects on salivary glands: dry mouth. Oral Dis. 2003 Jul;9(4):165-76. doi: 10.1034/j.1601-0825.2003.03967.x. PMID 12974516
- [Background] Rudolph JL. Antipsychotic (Non)selectivity: A Setup for Swallowing and Side-Effects in Seriously Ill Elderly Adults. J Am Geriatr Soc. 2017 Dec;65(12):2564-2565. doi: 10.1111/jgs.15168. Epub 2017 Nov 2. No abstract available. PMID 29095480
- [Background] Herzig SJ, LaSalvia MT, Naidus E, Rothberg MB, Zhou W, Gurwitz JH, Marcantonio ER. Antipsychotics and the Risk of Aspiration Pneumonia in Individuals Hospitalized for Nonpsychiatric Conditions: A Cohort Study. J Am Geriatr Soc. 2017 Dec;65(12):2580-2586. doi: 10.1111/jgs.15066. Epub 2017 Nov 2. PMID 29095482
- [Background] Keller H, Carrier N, Duizer L, Lengyel C, Slaughter S, Steele C. Making the most of mealtimes (M3): grounding mealtime interventions with a conceptual model. J Am Med Dir Assoc. 2014 Mar;15(3):158-161. doi: 10.1016/j.jamda.2013.12.001. No abstract available. PMID 24513225
- [Background] Gilmore-Bykovskyi AL, Rogus-Pulia N. Temporal Associations between Caregiving Approach, Behavioral Symptoms and Observable Indicators of Aspiration in Nursing Home Residents with Dementia. J Nutr Health Aging. 2018;22(3):400-406. doi: 10.1007/s12603-017-0943-y. PMID 29484354
- [Background] Chang CC, Roberts BL. Feeding difficulty in older adults with dementia. J Clin Nurs. 2008 Sep;17(17):2266-74. doi: 10.1111/j.1365-2702.2007.02275.x. PMID 18705703
- [Background] Serel Arslan S, Demir N, Karaduman AA. The Anxiety Level of Caregivers of Neurological Patients with Dysphagia. Dysphagia. 2017 Aug;32(4):570-574. doi: 10.1007/s00455-017-9801-7. Epub 2017 Apr 25. PMID 28444487
- [Background] Perneczky R, Wagenpfeil S, Komossa K, Grimmer T, Diehl J, Kurz A. Mapping scores onto stages: mini-mental state examination and clinical dementia rating. Am J Geriatr Psychiatry. 2006 Feb;14(2):139-44. doi: 10.1097/01.JGP.0000192478.82189.a8. PMID 16473978
- [Background] Kaiser BL, Thomas GR, Bowers BJ. A Case Study of Engaging Hard-to-Reach Participants in the Research Process: Community Advisors on Research Design and Strategies (CARDS)(R). Res Nurs Health. 2017 Feb;40(1):70-79. doi: 10.1002/nur.21753. Epub 2016 Sep 30. PMID 27686421
- [Background] Martin-Harris B, Brodsky MB, Michel Y, Castell DO, Schleicher M, Sandidge J, Maxwell R, Blair J. MBS measurement tool for swallow impairment--MBSImp: establishing a standard. Dysphagia. 2008 Dec;23(4):392-405. doi: 10.1007/s00455-008-9185-9. Epub 2008 Oct 15. PMID 18855050
- [Background] Morris JC. Clinical dementia rating: a reliable and valid diagnostic and staging measure for dementia of the Alzheimer type. Int Psychogeriatr. 1997;9 Suppl 1:173-6; discussion 177-8. doi: 10.1017/s1041610297004870. PMID 9447441
- [Background] Heller DA, Ahern FM, Pringle KE, Brown TV. Among older adults, the responsiveness of self-rated health to changes in Charlson comorbidity was moderated by age and baseline comorbidity. J Clin Epidemiol. 2009 Feb;62(2):177-87. doi: 10.1016/j.jclinepi.2008.05.009. Epub 2008 Aug 22. PMID 18722090
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Kayser-Jones J, Bird WF, Paul SM, Long L, Schell ES. An instrument to assess the oral health status of nursing home residents. Gerontologist. 1995 Dec;35(6):814-24. doi: 10.1093/geront/35.6.814. PMID 8557208
- [Background] Sahyoun NR, Lin CL, Krall E. Nutritional status of the older adult is associated with dentition status. J Am Diet Assoc. 2003 Jan;103(1):61-6. doi: 10.1053/jada.2003.50003. PMID 12525795
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Pearson WG Jr, Molfenter SM, Smith ZM, Steele CM. Image-based measurement of post-swallow residue: the normalized residue ratio scale. Dysphagia. 2013 Jun;28(2):167-77. doi: 10.1007/s00455-012-9426-9. Epub 2012 Oct 23. PMID 23089830
- [Background] McHorney CA, Robbins J, Lomax K, Rosenbek JC, Chignell K, Kramer AE, Bricker DE. The SWAL-QOL and SWAL-CARE outcomes tool for oropharyngeal dysphagia in adults: III. Documentation of reliability and validity. Dysphagia. 2002 Spring;17(2):97-114. doi: 10.1007/s00455-001-0109-1. PMID 11956835
- [Background] Navazesh M. Methods for collecting saliva. Ann N Y Acad Sci. 1993 Sep 20;694:72-7. doi: 10.1111/j.1749-6632.1993.tb18343.x. No abstract available. PMID 8215087
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] R Core Team. (2016). R: A Language and Environment for Statistical Computing. http://www.cran.rproject.org/package=ordinal/.
- [Background] Christensen RHB. (2015). Ordinal- Regression Models for Ordinal Data: R package version 2015.6-28.
- [Background] Bertrand F, Meyer N, & Maumy-Bertrand M. (2014). Partial Least Squares Regression for Generalized Linear Models: R package version 1.1.1.
- [Background] Steele CM, Bayley MT, Peladeau-Pigeon M, Nagy A, Namasivayam AM, Stokely SL, Wolkin T. A Randomized Trial Comparing Two Tongue-Pressure Resistance Training Protocols for Post-Stroke Dysphagia. Dysphagia. 2016 Jun;31(3):452-61. doi: 10.1007/s00455-016-9699-5. Epub 2016 Mar 2. PMID 26936446